CLINICAL TRIAL: NCT03980964
Title: Prospective Evaluation of Neuromuscular Electrical Stimulation (NMES) for Reducing Pain and Improving Functional Outcomes in Knee Osteoarthritis (OA) Patients
Brief Title: Evaluation of NMES for Reducing Pain and Improving Functional Outcomes in Knee OA Patients
Acronym: NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CyMedica Orthopedics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CY-0030-306
Record Dates: First submitted 2019-06-07; First posted 2019-06-10 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Knee Arthritis
Keywords: NMES; arthritis; knee pain; osteoarthritis; electrical stimulation therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: One-way crossover- Patients from the control cohort are allowed to crossover to the treatment cohort after 12 weeks of study enrollment, if a subject would request receiving knee intra-articular injections of hyaluronic acid (HA) or corticosteroids (CS) or opioids. Patients are also allowed to crossover to the treatment arm if they decide to drop out of the study due to the potential lack of clinical benefits from the sham treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active NMES (Experimental): Treatment arm receives an active NMES therapy including a conductive garment with NMES therapy, electrodes, and mobile app.
  Interventions: Device: Active NMES
- Inactive NMES (Sham Comparator): Control arm receives inactive NMES therapy including a conductive garment (no NMES and no electrodes), and mobile app.
  Interventions: Device: Active NMES

INTERVENTIONS:
Device: Active NMES — Daily home-based, mobile-app controlled, neuromuscular electrical stimulation (NMES) therapy

SUMMARY:
The present prospective trial is designed to evaluate the efficacy of CyMedica Orthopedics e-vive™ system, a multifunctional electrotherapy device providing neuromuscular electrical stimulation (NMES) for reducing pain and accelerating functional recovery in patients with knee osteoarthritis. This post-market trial will involve patients who have been diagnosed with knee osteoarthritis, Kelgren-Lawrence Grades II, III, and IV. It is hypothesized that the use of the CyMedica e-vive NMES can reduce pain, improve knee function, and improve quality of life.

DETAILED DESCRIPTION:
The study will be conducted at Lenox Hill Hospital, Northwell Health, located in New York, New York, and involve a total of 120 patients. All study patients will be evenly divided into two groups: (a) conductive garment and mobile app with NMES therapy; (b) conductive garment and mobile app without NMES therapy (sham).

Eligible patients will be evaluated according to the time and events schedule. Clinical outcomes will be assessed from 1 to 10 days before day of intervention and followed up after intervention over a 24 weeks ± 1 week study period.

These two groups will be analyzed using several outcome measures including validated patient-reported outcome measures including Visual Analogue Scale (VAS) pain level, the Knee Injury and Osteoarthritis Outcome Score (KOOS) JR., KOOS ADL, and WOMAC survey. Functional measures include isometric quadriceps strength, Time Up and Go (TUG), 6 minute walk test, repeated chair rise test, stair climb test, and number of steps recorded by an Apple Watch Series 3 or a Samsung watch. Reduction of use of anti-inflammatory medications (NSAIDS) and narcotics, use of ambulation assist devices, plan for TKA procedure survey, device compliance use, and patient satisfaction survey will be tracked The primary endpoint for the study is Visual Analogue Scale (VAS) pain The proprietary app for this product will be used to track device usage (intensity, duration of session, frequency of use), VAS, WOMAC, and KOOS JR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic Kellgren-Lawrence (KL) Grade 2, 3, or 4 OA by radiograph (AP tunnel view) within 30 days prior to day 0 visit, where the K-L grades are defined as:

   * Grade 0: no radiographic features of OA are present
   * Grade 1: doubtful joint space narrowing (JSN) and possible osteophytic lipping
   * Grade 2: definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph
   * Grade 3: multiple osteophytes, definite JSN, sclerosis, possible bony deformity
   * Grade 4: large osteophytes, marked JSN, severe sclerosis and definite bony deformity
2. Patients who are between the ages of 18 - 85 years
3. Patient has signed informed consent
4. Patient has access to a smartphone or tablet (Android or iOS)
5. Subject must be ambulatory.
6. Subject must be willing to stop taking any pain medications 24 hours prior any scheduled study visit.
7. Subjects must be proficient in English.
8. Subject must be willing and able to sign an informed consent document.
9. Subjects must be willing and able to comply with all study procedures for the duration of the clinical study.

Exclusion Criteria:

1. Subjects who have a body mass index > 40 at the time of consent. Exclusion of a patient with BMI>40 is up to the discretion of the PI.
2. Subjects with a diagnosis of inflammatory arthritis (rheumatoid arthritis, gout, joint infection, Lyme disease, SLE, etc.).
3. Subjects who have had an injury or an acute traumatic injury to the index knee within 6 months of screening will be excluded.
4. Subject must NOT have had arthroscopy within 8 weeks of randomization.
5. Subjects who have had treatment of the target knee with intra-articular injections of steroids within 8 weeks of screening.
6. Subjects who have had intra-articular injections of hyaluronic acid within 12 weeks of screening.
7. Subjects who have had a scheduled surgery on the target knee within the study period.

   (Note- Patients who are scheduled to go under surgery within the next 6 months will be excluded. Patients that are contemplating the surgery can be included.)
8. Subjects who have used electrotherapy or acupuncture for OA of the target knee within 4 weeks of screening
9. Subjects with significant and clinically evident mal-alignment of the target knee (> 10 degrees varus or valgus in the target knee).
10. Subjects with surgical metallic hardware in the target knee.
11. Subjects who have contraindications to MRI and X-rays, for example, implanted electrical devices (cardiac pacemakers, deep brain stimulators).
12. Subjects with a current malignancy or who have received treatment for malignancy with the last 5 years, with the exception of resected basal cell carcinoma and squamous cell carcinoma of the skin.
13. Subjects who have an active substance abuse problem (drugs or alcohol) or a history of chronic substance abuse (> 5 years).
14. Subjects with skin breakdown or infection in the area where the study device will be placed.
15. Subjects with any chronic conditions (e.g., diabetes, hypertension, congestive heart failure, etc.) that have not been well-controlled for at least 3 months prior to screening.
16. Subjects who have any ongoing litigation for worker's compensation.
17. Subjects with any condition, in the opinion of the Investigator that might interfere with the evaluation of the study objectives.
18. Subjects who are pregnant.
19. Subject must not have participated in a clinical study within the past 12 weeks that required the use of an investigational device, drug or biologic

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) pain level | 12 weeks post intervention
  Pain for a nominated activity causing the worst knee pain
Visual Analogue Scale (VAS) pain level | 12 weeks post intervention
  Worst pain at rest
Visual Analogue Scale (VAS) pain level | 12 weeks post intervention
  Worst pain walking

SECONDARY OUTCOMES:
Quadriceps strength | 12 weeks post intervention
  Isometric quadriceps strength or torque
TUG | 12 weeks post intervention
  Timed Up and Go test
Repeated chair rise | 12 weeks post intervention
  Repeated chair rise test
Stair climb | 12 weeks post intervention
  Stair climb
6 min walk test | 12 weeks post intervention
  6 min walk test
Activity | 12 weeks post intervention
  Average number of daily steps
Pain related medication | 12 weeks post intervention
  NSAIDS, Narcotics
Knee injections | 12 weeks post intervention
  HA and CS injections
Physical therapy | 12 weeks post intervention
  Utilization of physical therapy
Ambulation assist devices | 12 weeks post intervention
  Utilization of ambulation assist devices
Plan for TKA surgery | 12 weeks post intervention
  Plan for TKA surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No